CLINICAL TRIAL: NCT04844996
Title: Antilipidemic Ezetimibe Induces Regression of Endometriotic Explants in a Rat Model of Endometriosis
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Hakan Aytan, Professor Dr., Mersin University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 992903
Record Dates: First submitted 2021-04-10; First posted 2021-04-14 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Endometriosis
Keywords: endometriosis, ezetimibe, antilipidemics
MeSH Terms: conditions — Endometriosis | interventions — Pharmaceutical Preparations; Ezetimibe; Sodium Chloride; Organization and Administration

STUDY DESIGN:
Intervention Model Description: an experimental rat, randomized, drug versus placebo trial
Who Masked: Outcomes Assessor
Masking Description: the outcome assessors who measured the sizes of the post-treatment explants, and who histopathologically evaluated the explants were blinded to the groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ezetimibe group (Experimental): The endometriosis model was developed surgically in all 18 rats and pretreatment sizes of the endometriotic explants were measured. After randomization Ezetimibe (1 mg/kg/day (Ezetrol®, Merck Sharp Dohme, Istanbul, Turkey) was administered orally with gavage methodology to the 9 rats in the ezetimibe group for 28 days postoperatively.
  Interventions: Procedure: Surgical induction of endometriotic explants
- Control groups (Placebo Comparator): The endometriosis model was developed surgically in all 18 rats and pretreatment sizes of the endometriotic explants were measured. After randomization saline (1 ml/kg/day) was administered orally with gavage methodology to the 9 rats in the control group for 28 days postoperatively.
  Interventions: Procedure: Surgical induction of endometriotic explants

INTERVENTIONS:
Procedure: Surgical induction of endometriotic explants — Surgical induction of endometriosis was done as: A 5-cm vertical midline incision was made and a distal segment 1 cm in length of the right uterine horn was resected. The segment was split longitudinally, and a 5 X 5 mm piece was sectioned.
  This piece of uterine tissue was transplanted without removing the myometrium onto the inner surface of the right abdominal wall with the serosal surface apposed and secured with single nonabsorbable 5-0 polypropylene suture at the middle to the abdominal wall. The abdominal incision was closed in two layers
  Drug administration:
  Vehicle treatment (1 mL/kg/day saline) was administered orally to the control group with the gavage methodology. Ezetimibe (1 mg/kg/day (Ezetrol®, Merck Sharp Dohme, Istanbul, Turkey) was administered orally with gavage methodology to the rats in the study for 28 days postoperatively
  Other Names: Drug (ezetimibe 1mg/kg/day) and placebo (saline 1 ml/kg/day) administration

SUMMARY:
Current endometriosis therapy is based on interrupting the menstrual cycle and suppression of estrogen synthesis in order to induce atrophy of endometrial tissue. Progestins, oral contraceptives, androgenic agents, aromatase inhibitors, gonadotropin-releasing hormone analogues all play a role in the treatment of endometriosis. However, none of these treatments can definitely cure the disease and they require long-term use despite the side effects of the drug. It is clear that new treatment methods are needed for this disease, and therefore many different new treatment methods are being investigated. Some of the treatment methods have focused on inhibiting angiogenesis and inflammation, which seems to play an important role in the progression of the disease. In the present study, it was investigated whether ezetimibe which is a cholesterol absorption inhibitor with anti-inflammatory and antiangiogenic properties, has therapeutic effect on endometriosis in an experimental rat model.

DETAILED DESCRIPTION:
Endometriosis is a relatively common benign disorder that causes significant health problems with yet an unknown etiology. The disease which is defined as the presence of the endometrial gland and stroma outside the uterine cavity, was first described by the famous pathologist Von Rokitansky in 1860. Since then, new theories about the mechanism of its occurrence have been put forward, but no single theory has been holistic enough to explain all clinical presentations of the disease. Retrograde menstruation, stem cell theory, immune system, genetic and environmental factors are among the proposed theories. However, with the widespread use of molecular methods in recent years, more detailed information about its etiopathogenesis has been obtained and new approaches have been proposed for its diagnosis and treatment. Today, it is accepted that multiple factors, including ectopic endometrial tissue, altered immune system response, imbalanced cell proliferation and apoptosis, abnormal endocrine signal and genetic factors, play a role in the pathogenesis of endometriosis, which is a progressive, estrogen-dependent inflammatory disease.

In recent years, studies on the inflammatory and angiogenesis mechanisms that play a role in the pathogenesis of endometriosis have intensified in the treatment of the disease. Agents with anti-inflammatory and antiangiogenic effects have been experimentally shown to partially prevent the formation or reduce the size of endometriotic lesions in animal models. Statins like atorvastatin and simvastatin have been using in the treatment of coronary artery disease with their antilipidemic effects and are shown to have efficacy in animal endometriosis models with their anti-inflammatory and antiangiogenic properties.

Ezetimibe, which is a member of a different class of antilipidemic agents than statins, has similarly been shown to inhibit the release of substances that play a key role in the inflammatory process such as nuclear factor kappa, TNF-α and interleukin 1, and angiogenesis such as VEGF. With this mechanism of action, it may be hypothesized that this agent may have a possible therapeutic effect on endometriosis. Therefore in this study it was aimed to assess the potential therapeutic role of ezetimibe in the experimental rat endometriosis model.

ELIGIBILITY:
Inclusion Criteria:

* non-pregnant, sexually mature albino rats weighing between 180-240 g

Exclusion Criteria:

* pregnant, non-healthy, sexually immature, weighing <180 g

Ages: 3 Months to 12 Months | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
The volume of endometriotic explants in mm3. | 3 months
  The sizes of the explants were measured with a caliber. The spherical volume of each ectopic uterine tissue was calculated using the prolate ellipsoid formula (V [mm3] = 0.52 × width × length × height).
The amount of vascular endothelial growth factor | 5 months
  Immunohistochemical stains were performed with standard protocols. For immunohistochemical evaluation the intensity of the staining in each section was scored as intense (++++), moderate (+++), mild (++), and none (+).
The amount of tumor necrosis factor alpha | 5 months
  Immunohistochemical stains were performed with standard protocols. For immunohistochemical evaluation the intensity of the staining in each section was scored as intense (++++), moderate (+++), mild (++), and none (+).
The number of mast cells | 5 months
  The number of the mast cells stained with toluidine blue was counted under x20 magnification separetely in 5 different areas of the endometrium, myometrium and perimetrium in each specimen (15 different areas in each subject).

CONTACTS AND LOCATIONS:
Locations (1):
- Mersin University, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No